CLINICAL TRIAL: NCT02759783
Title: A Randomised Trial of Conventional Care Versus Radioablation (Stereotactic Body Radiotherapy) for Extracranial Oligometastases
Brief Title: Conventional Care Versus Radioablation (Stereotactic Body Radiotherapy) for Extracranial Oligometastases
Acronym: CORE
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Institute of Cancer Research, United Kingdom (Other); National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR4323; 182152 (Other: IRAS); ISRCTN45961438 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2016-04-26; First posted 2016-05-03 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Prostate Cancer; Breast Cancer; Carcinoma, Non-Small-Cell Lung
Keywords: Radiotherapy; oligometastases; SBRT
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (Active Comparator): Standard of care (SOC) is at the discretion of the local oncologist.
  Interventions: Other: Standard of Care
- Standard of Care + SBRT (Experimental): Patients randomised to SBRT will receive a dose and fractionation regimen dependent on the metastatic site and proximity to normal tissues. If allocated to SBRT, SBRT will precede SOC.
  Interventions: Radiation: SBRT; Other: Standard of Care

INTERVENTIONS:
Radiation: SBRT — Patients will receive a dose and fractionation regimen dependent on the metastatic site and proximity to normal tissues. If allocated to SBRT, SBRT will precede SOC. All patients should commence SOC therapy within 4 weeks of completing SBRT treatment.
  Other Names: Stereotactic body Radiotherapy; SABR
  Arms: Standard of Care + SBRT
Other: Standard of Care — Choice of standard of care treatment at the discretion of the local oncologist. This may include: Chemotherapy, Endocrine therapy, surgery, palliative radiotherapy

SUMMARY:
Metastatic spread of cancer from its primary site to distant organs is the commonest cause of death from cancer. The term oligometastases describes an intermediate metastatic state, in which cancer exists as a limited number of metastases at first, before cells acquire the ability to metastasise more widely. For the large majority of solid cancers, once metastatic disease has been diagnosed the chances of cure are small. There are several situations where this is not the case, but it is not known if stereotactic body radiotherapy (SBRT) for oligometastatic disease will alter outcomes or whether the toxicity burden of this treatment is justified. SBRT is targeted radiotherapy which destroys cancer cells in the area of the body it is aimed at however low dose radiation may be received by surrounding tissue.

It is difficult to quantify incidence of patients with multiple primary cancers developing at intervals that are representative of oligometastatic stage IV disease, (defined for the purposes of this trial as ≤ 3 metastatic sites). However an increase in the use of surveillance imaging, together with improved diagnostic sensitivity has led to the diagnosis of patients with asymptomatic oligometastatic relapse becoming a more common clinical occurrence. The CORE study is a randomized controlled trial that will be conducted in patients with cancer in one of three primary sites where oligometastatic disease relapse is a common clinical scenario: breast, prostate and non-small cell lung cancer (NSCLC). The study will evaluate the use of SBRT in this patient population.

Eligible patients who consent to participate in this clinical trial will be randomized to receive standard care or standard care plus SBRT we hope to recruit approximately 206 patients to the study and the primary outcome measure is progression free survival.

DETAILED DESCRIPTION:
CORE is a phase II/III, multi-centre, non-blinded, parallel group randomised controlled trial in patients with breast, prostate or NSCLC primary cancer comparing standard of care (SOC) with or without SBRT for extra-cranial metastases. The aim of the phase II study is to demonstrate 1) feasibility of recruitment, 2) deliverability of the study in a multi-centre setting and 3) activity of SBRT, based on progression free survival, across the three tumour types. If all three aims are achieved the trial will be amended to roll into parallel tumour-site specific phase III trials.

Eligible patients are those with either primary breast, prostate or NSCLC who have presented with ≤3 extra-cranial, metachronous, oligometastases, all suitable for SBRT. Patients will be randomised in a 1:1 ratio to either SOC or SOC with the addition of SBRT. Choice of SOC treatment is at the discretion of the local oncologist and defined per patient prior to randomisation (see section 8). Patients randomised to SBRT+SOC will receive a dose and fractionation regimen dependent on the metastatic site and proximity to dose limiting organs and normal tissues. Treatment will take place within 6 weeks of randomisation. The average scheme would be 3 treatments over 5 days but the maximum period of SBRT duration could be 8 treatments over 19 days.

All patients will be reviewed every 3 months with a clinical examination and tumour markers (where applicable) during years 1 and 2, and 6 monthly thereafter to 5 years. Staging and follow up imaging protocols will be tumour type dependent:

* Breast: 3 monthly CT scans for years 1 and 2, and 6 monthly thereafter to 5 years.
* NSCLC: 3 monthly CT scans for years 1 and 2, 6 monthly to year 3, then annually to 5 years.
* Prostate: CT scans will be performed at 6, 12 and 24 months with imaging triggered by appropriate PSA rises. A rising PSA defined as 2 successive PSA rises from nadir, measured a minimum of 4 weeks apart. If the overall PSA rise has a doubling time of ≥ 3 months or the PSA level has doubled the original PSA value at trial entry or if clinically indicated, then restaging should be considered.

All patients will have a toxicity assessment at each clinic visit and patient reported quality of life (QOL) assessment at 3, 6, 12, 18 and 24 months.

ELIGIBILITY:
Inclusion criteria

1. Age ≥ 18 years
2. WHO performance status 0-2
3. Histological confirmation of primary malignancy (histological confirmation of metastasis is not mandatory but should be performed in any situation where there is diagnostic uncertainty). Patients with breast, NSCLC or prostate primary malignancies are eligible.
4. Predicted life expectancy > 6 months
5. ≤ 3 metastatic lesions (total). A maximum of 2 different organ systems (e.g. liver, lung, bone, nodal) may contain metastases but the total number of lesions must not exceed 3. For example, a patient with 3 liver metastases or 1 liver metastasis and 2 lung metastases would be eligible. A patient with 1 lung metastasis, 1 liver metastasis and an adrenal metastasis is ineligible.
6. All metastases must be visible, imaging defined targets and be suitable for treatment with SBRT in accordance with the dose fractionation options specified in the protocol. (See the associated CORE trial radiotherapy delivery guidelines for detailed SBRT guidance by metastatic site)
7. Patients who have received prior ablative therapy (e.g. surgery, RFA or SBRT) for metastatic disease are eligible, as long as this site is controlled on imaging at the point of trial entry and the total number of metastases over time since diagnosis of metastatic disease does not exceed 3. Patients with 2 or 3 metastases in which ablative therapy (e.g. surgery/RFA) to 1 site is deemed appropriate as part of standard therapy may be entered into the trial following successful delivery of the ablative treatment. Ablative therapy (e.g. surgery, RFA, cryoablation, SBRT) is not permissible as a standard of care option following randomisation for patients as part of the trial.
8. Only patients with metachronous metastatic disease presentation are eligible. Primary site must be controlled.

   NSCLC patients with synchronous presentation of a single brain metastasis with the primary lung malignancy are eligible as long as both sites of disease have received radical treatment. Both primary lung site and solitary synchronous brain metastasis must be controlled at trial entry, and the total number of metastases over time including the brain metastasis must not exceed 3.

   Permissible disease-free intervals are:

   Breast: ≥ 6 months from completion of radical treatment including any adjuvant therapy to diagnosis of metastases. Patients who have relapsed whilst on adjuvant endocrine therapy are eligible.

   NSCLC: ≥ 4 months from completion of radical treatment (not including any adjuvant chemotherapy) to diagnosis of metastases.

   Prostate: ≥ 6 months from completion of radical treatment including any adjuvant therapy to diagnosis of metastases. Patients who have relapsed whilst on adjuvant endocrine therapy are eligible.
9. Only patients who are systemic therapy naïve in the metastatic setting are eligible. Prior systemic therapy in the adjuvant setting is permitted. Patients who have had a change in endocrine therapy due to the diagnosis of oligometastatic disease can be entered into the CORE trial as long as entry is within 8 weeks of this change in therapy for prostate cancer patients and within 10 weeks of this change in therapy for breast cancer patients.
10. Adequate baseline organ function to allow SBRT to all relevant targets dependent on location of metastatic subsite
11. Negative pregnancy test (for women of childbearing potential)
12. Written informed consent.

Exclusion criteria

1. Intra-cranial metastases (not meeting above inclusion criterion 8).
2. Malignant pleural effusion
3. Malignant peritoneal disease
4. Any single metastasis >6cm,( >5cm for lung metastases)
5. Prior radiotherapy to a site that precludes safe delivery of SBRT
6. Co-morbidities precluding staging or follow up imaging, or precluding procedures required to facilitate SBRT
7. Loco-regional nodal relapse where surgery is considered the standard of care and is technically feasible. Patients with internal mammary chain or supraclavicular fossa lymph node relapses of breast cancer are eligible if SBRT dose constraints can be met. Patients with axillary nodal relapse from breast cancer are excluded
8. Spinal cord compression, or impingement of the cord or any other situation whereby the clinician feels that urgent radiotherapy to the spine is required (within 24 hours)
9. Any condition or significant clinical co-morbidities that preclude the safe delivery of SBRT (e.g. history of clinically significant diffuse interstitial lung disease if SBRT to lung metastases or lesions adjacent to lungs are considered or clinically significant colitis i.e. ulcerative colitis /Crohn's disease if SBRT to the pelvis or abdomen is considered).
10. Prostate cancer patients who have relapsed on Androgen Deprivation Therapy (ADT) which was started for biochemical relapse without staging investigations to define their relapse status, or who have relapsed on CAB which was started for biochemical relapse.
11. Prostate cancer patients receiving or have previously received abiraterone, enzalutamide or chemotherapy e.g. docetaxel.
12. Previous malignancy within the last 2 years (except basal cell carcinoma or squamous cell carcinoma of the skin), or if previous malignancy is expected to significantly compromise 5 year survival.
13. Patients whose entry to the trial will cause unacceptable clinical delays to their planned management.
14. Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 60 months post treatment
  Time from randomisation to evidence of progression of cancer at any site or death from any cause

SECONDARY OUTCOMES:
Feasibility of recruitment | 3 years from first patient
  Recruitment rate and proportion of patients receiving SBRT (if allocated) in the absence of new developing widespread disease
Feasibility of SBRT delivery | 3 years from first patient
  Recruitment of patients receiving SBRT within the dosimetric constraints
Overall Survival | 60 months post treatment
  Time from randomisation until time of death from any cause
Local lesion control | 60 months post treatment
  Time from randomisation until radiological evidence of progression at the treated site and be measured on a lesion based on analysis using RECIST criteria.
Clinical reported acute and late toxicity | 60 months post treatment
  Clinician reported acute and late toxicity will be graded using NCI CTCAE v4.0 / RTOG systems. Acute events are defined as those occurring up to 3 months follow-up; late events are reported from 6 months post randomisation.
Patient reported Quality of Life | Pre-treatment and at 3,6,12,18 and 24 months post treatment
  Patient reported quality of life will be measured using EORTC QLQ C30

OTHER OUTCOMES:
Freedom from widespread metastatic disease (FFWMD) | Pre-treatment and at 3,6,9,12,15,18,21,24,30,36,42,48,54 and 60 months post treatment
  FFWMD will be measured from the time of randomisation until radiological evidence of disease progression, which is not suitable for radical salvage therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Khoo, MD, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (30):
- Australia (9):
  - Liverpool Hospital, Liverpool, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - GenesisCare - Adelaide Radiotherapy Centre, Adelaide, South Australia
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Austin Health, Melbourne, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- United Kingdom (21):
  - Churchill Hospital, Oxford, Oxfordshire
  - Mount Vernon Cancer Centre, London, Surrey
  - Belfast City Hospital, Belfast
  - Queen Elizabeth Hospital, Birmingham
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrooke's Hospital, Cambridge
  - The Beatson, Glasgow
  - Royal Surrey County Hospital, Guildford
  - St James's University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Royal Marsden Hospital, London
  - Guy's Hospital, London
  - St Bartholomew's Hospital, London
  - University College Hospital, London
  - The Christie Hospital, Manchester
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - James Cook University Hospital, Middlesbrough
  - Freeman Hospital, Newcastle upon Tyne
  - Nottingham City Hospital, Nottingham
  - Weston Park Hospital, Sheffield
  - Royal Marsden Hospital, Sutton